CLINICAL TRIAL: NCT00235183
Title: Plasma Transfusion in Liver Transplantation : a Randomized, Double Blind, Multicenter Trial of Methylene Blue, Solvent/Detergent and Quarantined Plasma.
Brief Title: Plasma Transfusion in Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFS plasma trial
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Bleeding in Liver Transplantation
Keywords: plasma; bleeding; liver transplantation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Quarantined FFP (Active Comparator): Quarantined FFP
  Interventions: Other: plasma
- Methylene blue FFP (Active Comparator): Methylene blue FFP
  Interventions: Other: plasma
- Solvent detergent FFP (Active Comparator): Solvent detergent FFP
  Interventions: Other: plasma

INTERVENTIONS:
Other: plasma — transfusion of more than 15 mL/Kg of plasma

SUMMARY:
The aim of the study is to compare the clinical efficacy of three types of plasma secured on the viral level either by quarantine or by chemical treatment in patients undergoing liver transplantation.

DETAILED DESCRIPTION:
Three types of plasma are transfused in bleeding patients undergoing liver transplantation:

* quarantined plasma,
* methylene blue treated plasma,
* solvent/detergent plasma. The main purpose is to show that the volume of methylene blue treated plasma consumed intraoperatively is equivalent to that of the 2 other types of plasma.

In addition, the correction of coagulation abnormalities are studied.

ELIGIBILITY:
Inclusion Criteria:

* age 18 yo and above
* consent is signed,
* liver transplantation is indicated,
* plasma is transfused

Exclusion Criteria:

* multiorgan transplantation (except combined kidney and liver transplantation)
* allergy to methylene blue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Volume of transfused plasma during surgery | 5 years

SECONDARY OUTCOMES:
correction of coagulation abnormalities | 5 years
immediate and delayed adverse events | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Yves Ozier, MD, PhD, Principal Investigator — Hôpital Cochin, Paris, France; Emmanuel Samain, MD, PhD, Principal Investigator — hôpital Jean Minjoz, Besançon, France; Marie - Christine Gillon, MD, Principal Investigator — Hôpital Paul Brousse, Villejuif, France; Loïc Villalon, MD, Principal Investigator — Hôpital Pontchaillou
Locations (1):
- EFS, Paris, France

REFERENCES:
- [Derived] Bartelmaos T, Chabanel A, Leger J, Villalon L, Gillon MC, Rouget C, Gomola A, Denninger MH, Tardivel R, Naegelen C, Courtois F, Bardiaux L, Giraudeau B, Ozier Y. Plasma transfusion in liver transplantation: a randomized, double-blind, multicenter clinical comparison of three virally secured plasmas. Transfusion. 2013 Jun;53(6):1335-45. doi: 10.1111/j.1537-2995.2012.03895.x. Epub 2012 Sep 24. PMID 22998014